CLINICAL TRIAL: NCT04406766
Title: Evaluation of a Data Transmission Solution for Connected Nutrition Pump for Patients Treated by Home Parenteral Nutrition (HPN). Proof of Concept, Prospective, Monocentric, Non-randomized, and Open-label Study.
Brief Title: Evaluation of a Connected Parenteral Pump for Patients Treated by Home Parenteral Nutrition (HPN).
Acronym: SERENE-eNUTRI
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Context of the COVID-19 pandemic, strict eligibility criteria (especially 15 km radius from the CHUGA) significantly reducing the active file and the recruitment capacities.
Sponsor: University Hospital, Grenoble (Other)
Collaborators: Clinical Investigation Centre for Innovative Technology Network (Network); MAATEL (Unknown); Orange Labs (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: 38RC19.343
Record Dates: First submitted 2020-05-22; First posted 2020-05-28 (Actual); Last update posted 2023-01-09 (Actual); Status verified 2021-01

CONDITIONS: Parenteral Nutrition, Home
Keywords: Connected feeding pump; Reduction of costs due to late management of complications; Patients quality of life improvement; Clinical management of patients' pathology improvement
MeSH Terms: conditions — Hyperphagia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Connected nutrition pump system (Experimental)
  Interventions: Device: Connected nutrition pump system

INTERVENTIONS:
Device: Connected nutrition pump system — For the patient, it consists of the installation of the connected pump at his home for a duration of one month.
  Infusion data and events will be continuously collected and transmitted by the 4 different modes (LoRaAN, BLE , GSM and multimodality).Transmitted data won't be used to change the follow up of the patient.
  At the end of the month, patients will be solicited by an ergonomic engineer to complete a specific questionnaire in order to evaluate the future acceptability of the proposed solution.

SUMMARY:
Patients requiring long-term home parenteral nutrition (HPN) suffer from chronic intestinal insufficiency. The causes of this syndrome can be either anatomical (extensive resection of the small bowel) or functional (occlusion, pseudo-occlusion, malabsorption). Consequences mean that patients are unable to cover their oral energy and / or hydroelectrolytic needs.

As a result, these patients survive only through a nutritional support by the venous route (parenteral nutrition). However, this lifesaving therapy requires complex technological nutritional support issues at home, which will influence the personal life of the patients.

At home, HPN therapy is performed by nutrition pumps providing a constant flow and able to detect anomalies.

In this context, the development of connected systems that allow informations transmission could help patient's caregiving by the different persons involved in his follow-up (prescribing physicians, home support nurses, patients and relatives, manufacturers).

The main objective of this study is to evaluate the performance of an end-to-end data transmission chain which integrates a nutrition pump connected to a medical IoT module (developped by Maatel) able to send information to an applicative layer (software interface PatHView2, developped by Orange Labs) via different transmission modes : LoRaWAN (Long Range Wide-area network), BLE (Bluetooth Low Energy), GSM LTE-M (Global System for Mobile Communications, Long Term Evolution - Machine Type Communication).

ELIGIBILITY:
Inclusion Criteria:

* Age < 18 years
* Patient receiving a home parenteral nutrition (HPN) and followed by the Artificial Nutrition Service of the CHUGA
* Patient carrying out all his infusions at home during the month of use of the connected pump (constraint due to the LoRaWAn transmission mode)
* Patient affiliated to the French social security system or an equivalent system
* Patient who has signed consent form

Exclusion Criteria:

* Presenting any other pathology or treatment that the physician may deem incompatible with this study
* Patient under exclusion period from another study
* Protected persons (patient concerned by articles L1121-5, L1121-6, L1121-8 of the French public health code)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2020-09-28 (Actual); Primary Completion 2021-07-16 (Actual); Study Completion 2021-07-16 (Actual)

PRIMARY OUTCOMES:
Ratio of all data and anomaly events correctly transmitted from the connected infusion pump to the software interface. | 1 month
  Evaluate the ratio of data (volume administered with the perfusion cycles over 24 hours; duration, velocity rate and mode of the perfusions) and events (occlusion of the venous route and presence of bubble in the infusion line) correctly transmitted in different transmission modalities (LoRaWan, BLE+GSM, GSM LTE-M, multimodality) from the connected infusion pump to the software interface.

SECONDARY OUTCOMES:
Volume of all data and anomaly events correctly transmitted from the nutrition pump to the software interface, compared to the volume of data to be transmitted. | 1 month
  Evaluate the ratio of all data (volume administered with the perfusion cycles over 24 hours; duration, velocity rate and mode of the perfusions) and events (occlusion of the venous route and presence of bubble in the infusion line) correctly transmitted in terms of volume using different transmission modalities (LoRaWan, BLE+GSM, GSM LTE-M, multimodality), from the connected infusion pump to the software interface.
Type and variable (value / field / date / time) for data and events from extracted files : - from the pump before the IoT module; - from the software interface. | 1 month
  Evaluate the ratio of each data type (volume administered with the perfusion cycles over 24 hours; duration, velocity rate and mode of the perfusions) and events (technical notifications of system use) correctly transmitted through the four transmission modalities (LoRaWan, BLE+GSM, GSM LTE-M, multimodality), from the connected infusion pump to the software interface. This target will be verified if the proportion of the main target is < 98%.
Frequency and typology of problems encountered. | 1 month
  Descriptive analysis of the problems encountered.
- Quantitative evaluation: number of cases in which the physician would have changed the patient follow-up over the entire study ; - Qualitative evaluation: nature of the follow-up change (no change, delayed change, immediate change). | 1 month
  Quantitative and qualitative evaluation of the proposed solution (software interface) in terms of medical reasoning help on the potential improvement of patient follow-up (i.e. compliance with a prescription).
Analysis of the efficacy, the efficiency, the difficulties and usage errors of the software interface by the medical team according to specific scenarios tests performed with an ergonomist (with voice and screen recording). | 1 month
  Evaluate the usability of the software interface by the medical team (physicians, nurses, ...).
Customised hetero-questionnaire at the end study visit. | 1 month
  Assess the acceptability of the proposed solution (connected pump) by the patient.

CONTACTS AND LOCATIONS:
Overall Officials: Eric Fontaine, MD, Principal Investigator — CHU Grenoble Alpes
Locations (1):
- CHU Grenoble Alpes, Grenoble, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Pironi L, Miglioli M, Ruggeri E, Longo N, Suriani U, Maselli S, Gnudi S, Barbara L. Home parenteral nutrition for the management of chronic intestinal failure: a 34 patient-year experience. Ital J Gastroenterol. 1993 Oct;25(8):411-8. PMID 8286774
- [Background] Detsky AS, McLaughlin JR, Abrams HB, L'Abbe KA, Whitwell J, Bombardier C, Jeejeebhoy KN. Quality of life of patients on long-term total parenteral nutrition at home. J Gen Intern Med. 1986 Jan-Feb;1(1):26-33. doi: 10.1007/BF02596321. PMID 3095514
- See also: Related Info — https://maatel.com/savoir-faire/etudes-de-cas-conception-electronique/serene-iot/
- See also: Related Info — https://www.has-sante.fr/upload/docs/application/pdf/2008-07/rapport_nutrition_parenterale_a_domicile_2008-07-31_14-29-41_874.pdf